CLINICAL TRIAL: NCT05436496
Title: CD19/70 Bi-specific CAR-T Cells Targeting B Cell Malignancies
Brief Title: CD19/70 Bi-specific CAR-T Cell Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-22008
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: B Cell Malignancies
Keywords: CAR-T; B cell Malignancies; CD19; CD70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bi-4SCAR-CD19/70 T Cell Therapy for CD19 and/or CD70 positive B cell malignancies (Experimental)
  Interventions: Biological: bi-4SCAR CD19/70 T cells

INTERVENTIONS:
Biological: bi-4SCAR CD19/70 T cells — Infusion of bi-4SCAR CD19/70 T cells at 10^6 cells/kg body weight via IV

SUMMARY:
The purpose of this study is to assess the feasibility, safety and efficacy of CD19/70 bi-specific CAR-T cell therapy in patients with CD19 and/or CD70 positive B cell malignancies. Another goal of the study is to learn more about the safety and function of the anti-CD19/70 bi-specific CAR-T cells and their persistency in patients.

DETAILED DESCRIPTION:
Patients with refractory and/or recurrent B cell malignancies have poor prognosis despite complex multimodal therapy. Despite impressive progress, more than 50% of patients treated with CD19-targeting chimeric antigen receptor T cells (CAR19) experience progressive disease. Further, more than 40% patients with progressive large B cell lymphoma (LBCL) experienced reduced or lost expression of CD19 on the tumor cells after CAR19 treatment; low surface CD19 density before treatment was associated with progressive disease. Therefore, novel curative approaches are needed. The investigation attempts to use genetically modified T cells to express a 4th generation lentiviral anti-CD19/70 bi-specific CAR (bi-4SCAR-CD19/70). The CAR molecules enable the T cells to recognize and kill tumor cells through the recognition of a surface antigen, CD19 or CD70, which is expressed at high levels on tumor cells but not at significant levels on normal tissues.

CD70 is highly expressed in many cancers, but limited in normal tissues, it is a potential CAR-T therapeutic target. Expression of CD70 was observed on multiple tumor types including solid tumor as well as B cell malignancies. In addition, it has been reported that anti-CD70 CAR T-cells can eliminate CD70-positive cells and exhibit strong anti-tumor effects in preclinical animal models. The CD70 targeted CAR-T cells with binding moiety of CD70 specific scFv exhibited a higher affinity and antitumor effect against CD70-positive tumor cells. A potential strategy to prevent relapse due to antigen escape is to infuse T-cells capable of recognizing multiple antigens.

To overcome tumor escape of single target antigen and enhance in vivo CAR-T efficacy, a novel bi-specific CD19/70 CAR-T therapy regimen is developed to include booster and consolidation CAR-T applications to target highly-refractory B cell cancer. The aim is to evaluate safety and long term efficacy of the bi-CAR-T therapy strategy in CD19 and/or CD70 positive cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 6 months.
2. malignant B cell surface expression of CD19 or CD70 molecules.
3. the KPS score over 80 points, and survival time is more than 1 month.
4. greater than Hgb 80 g/L.
5. no contraindications to blood cell collection.

Exclusion Criteria:

1. accompanied with other active diseases and difficult to assess patient response.
2. bacterial, fungal, or viral infection, unable to control.
3. living with HIV.
4. active HBV or HCV infection.
5. pregnant and nursing mothers.
6. under systemic steroid treatment within a week of the treatment.
7. prior failed CD19 and CD70 CAR-T treatment.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety of fourth generation bi-4SCARCD19/70 T cells in patients with B cell malignancies | 12 weeks
  Safety of fourth generation bi-4SCARCD19/70 T cells in patients with B cell malignancies using CTCAE 4 standard to evaluate the level of adverse events standard to evaluate the level of adverse events

SECONDARY OUTCOMES:
Anti-tumor activity of fourth generation bi-4SCARCD19/70 T cells in patients with relapsed or refractory B cell malignancies | 1 year
  Scale of CAR copies (for efficacy)
Anti-tumor activity of fourth generation bi-4SCARCD19/70 T cells in patients with relapsed or refractory B cell malignancies | 1 year
  Scale of leukemic cell burden (for efficacy)

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No